CLINICAL TRIAL: NCT06836752
Title: A Randomised, Open Label, Controlled, Parallel-group Study to Explore the Effects of 24 Weeks Intake of Yoghurt on Glucose Metabolism in Subjects at High Risk of Type 2 Diabetes Mellitus
Brief Title: Effects of Yoghurt Consumption on Glucose Metabolism in Prediabetic Subjects
Acronym: SNOWFALL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The current operational setting is not sustainable and very unlikely to deliver the planned enrollment of 60 participants. Even with significant protocol amendments, these challenges would remain.
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 23REX0060026
Record Dates: First submitted 2025-01-13; First posted 2025-02-20 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Prediabetes
Keywords: Randomized controlled trial; Prediabetes
MeSH Terms: conditions — Prediabetic State | interventions — Yogurt; Milk

STUDY DESIGN:
Intervention Model Description: Randomised, open label, controlled, parallel-group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yoghurt (Experimental): 2% fat yoghurt. Subjects will consume two servings (125 g/serving) of the test product per day.
  Interventions: Other: Yoghurt
- Milk (Placebo Comparator): 2% fat cow's milk. Subjects will consume two servings (125 g/serving) of the control product per day.
  Interventions: Other: Milk

INTERVENTIONS:
Other: Yoghurt — 250 g per day
  Arms: Yoghurt
Other: Milk — 250 g per day
  Arms: Milk

SUMMARY:
The purpose of this study is to explore the effects of yoghurt consumption on glucose metabolism in prediabetic subjects.

DETAILED DESCRIPTION:
Study population: the study population will consist of 60 (30 per group) subjects (men and women) at high risk of type 2 diabetes mellitus (T2DM), aged 18-65 years (inclusive), body mass index (BMI) 25.0 (inclusive) - 35.0 kg/m2 (exclusive), diagnosed with prediabetes, defined as fasting plasma glucose levels 100-125 mg/dL (5.6-6.9 mmol/L) (inclusive), randomised in a test and control group.

Intervention comprises of two study periods: a refrain period from dairy products and pro-, pre- and synbiotic supplements in any form, for 2 weeks, followed by an intervention period of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Signed ICF
2. Male/Female 18-65 years
3. BMI 25-35 kg/m2
4. FPG 100-125 mg/dL
5. At least one relative with T2DM
6. BW maintained (<3%)
7. Female postmenopausal or sterile or using contraceptive method
8. Ability to comply with study protocol form
9. Access to a refrigerator at home for study products storage
10. Ability to collect and store stool samples
11. Coverage by French health insurance
12. Agreement to be registered in the national database of subjects participating in clinical research
13. Ability to complete ePRO
14. FPG 100-125 mg/dL at randomisation visit

Exclusion Criteria:

1. Diagnosis of T2DM, T1DM, or on antidiabetic medications
2. Medications or supplements affecting gut microbiota or causing hyperglycemia
3. Systemic antibiotic treatment
4. Treatment interfering with BW and bariatric surgery
5. Liver, renal, cardiovascular, respiratory, endocrine, metabolic disorders, or iatrogenic immunodeficiency
6. Chronic gastro-intestinal disorders or recent use of laxatives
7. Recent surgery or general anesthesia
8. Donation/Loss of blood
9. Inability to comply with dietary restriction
10. Allergy or intolerance to study product ingredients
11. Excessive consumption of alcohol
12. Smoker
13. Pregnancy, breast-feeding or change in contraceptive methods
14. Situation interfering with optimal participation
15. Participation in other clinical study
16. Living in the same home as another participant
17. Employees, family members of Danone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2025-09-16 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Change in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) calculated as fasting serum insulin (FSI) levels (mU/L) multiplied by fasting plasma glucose (FPG) levels (mmol/L) divided by 22.5. | Change from Baseline to Week 24
Change in FPG [mmol/L] | Change from Baseline to Week 24
Change in 2-h post load Glucose Area Under the Curve (AUC) [mmol/L· min] measured during 2-hour oral glucose tolerance test (OGTT) | Change from Baseline to Week 24

SECONDARY OUTCOMES:
Change in Body Weight [kg] | Change from Baseline to Week 12 and to Week 24
Change in Body Mass Index (BMI) [kg/m²] as calculated by body weight (kg) divided by square of height (m) | Change from Baseline to Week 12 and to Week 24
Change in Waist Circumference [cm] | Change from Baseline to Week 12 and to Week 24
Change in Fat Mass as measured by Bioelectrical Impedance Analysis (BIA) [kg] | Change from Baseline to Week 24
Change in Fat Mass Percentage as measured by BIA (%) | Change from Baseline to Week 24
Change in Visceral Adipose Tissue mass [g] as measured by BIA [g] | Change from Baseline to Week 24
Change in Fat Free Mass as measured by BIA [kg] | Change from Baseline to Week 24
Change in fasting plasma Glycated Haemoglobin A1c (HbA1C) [%] | Change from Baseline to Week 12 and to Week 24
Change in FSI levels [mU/L] | Change from Baseline to Week 12 and to Week 24
Change in HOMA-IR calculated as FSI (mU/L) multiplied by FPG, (mmol/L) divided by 22.5 | Change from Baseline to Week 12
Change in FPG levels [mmol/L] | Change from Baseline to Week 12
Change in Glucose tolerance as measured by plasma glucose at 30-, 60-, and 120-min post load during 2-hour OGTT [mmol/L] | Change from Baseline to Week 24
Change in Insulin secretion as measured by serum insulin at 30-, 60-, and 120-min post load during 2-hour OGTT [mU/L] | Change from Baseline to Week 24
Change in β-cell function as measured by Homeostatic Model Assessment of β-cell function (HOMA-β) calculated as follows: 20 x FSI levels (mU/L) divided by FPG levels (mmol/L) subtracted by 3.5 | Change from Baseline to Week 24
Change in β-cell response as measured by Insulinogenic index (IGI), calculated from the OGTT as delta serum insulin (0-30 min) (µU/mL) divided by delta plasma glucose (0-30 min) (mg/dL) | Change from Baseline to Week 24
Change in whole-body insulin sensitivity as measured by Matsuda index, calculated from the OGTT as follows: (10,000/square root of (FPG (mg/dL) x FSI (mU/L)) x (mean plasma glucose (mg/dL) x mean serum insulin (mU/L) during OGTT]) | Change from Baseline to Week 24
Change in Disposition Index (DI), a composite marker of first phase insulin secretion and insulin sensitivity calculated from the OGTT as follows: Matsuda index * [AUC30min serum insulin (pmol/L) / AUC30min plasma glucose (mmol/L)], where AUC30min is the | Change from Baseline to Week 24
Change in Muscle Insulin Sensitivity Index (MISI), calculated from the OGTT as the slope of the least square fit to the decline in plasma glucose concentration (mmol/L) from peak to nadir divided by the mean serum insulin (pmol/L) during OGTT | Change from Baseline to Week 24
Change in Hepatic Insulin Resistance Index (HIRI) calculated from the OGTT as follows: the product of the plasma glucose (mmol/L) area under the curve and serum insulin (pmol/L) area under the curve during the first 30min of the OGTT | Change from Baseline to Week 24
Change in fasting circulating concentrations of alpha-hydroxyisocaproic acid (HICA), alpha-hydroxyisovaleric acid (HIVA) and alpha-hydroxy-beta-methylvaleric acid (HMVA) (μmol/L) | Change from Baseline to Week 24
Change in plasma Alanine Aminotransferase (ALAT) [U/L]) | Change from Baseline to Week 12 and to Week 24
Change in plasma Aspartate Aminotransferase (ASAT) [U/L]) | Change from Baseline to Week 12 and to Week 24
Change in Fibrosis 4 index (FIB-4) calculated as (Age (years) x ASAT (U/L) / (Platelets (109/L) x square root of ALAT (U/L))) | Change from Baseline to Week 12 and to Week 24
Change in fasting serum Total Cholesterol (TC) [mmol/L] | Change from Baseline to Week 12 and to Week 24
Change in fasting serum High Density Lipoprotein (HDL) [mmol/L] | Change from Baseline to Week 12 and to Week 24
Change in fasting serum Low Density Lipoprotein (LDL) [mmol/L] | Change from Baseline to Week 12 and to Week 24
Change in fasting serum Triglycerides (TG) [mmol/L] | Change from Baseline to Week 12 and to Week 24
Change in Energy intake from 3 non-consecutives days of 24-h dietary recalls [kcal/day] | Change from Baseline to Week 12 and to Week 24
Change in macronutrients intake from 3 non-consecutives days of 24-h dietary recalls [g/day] | Change from Baseline to Week 12 and to Week 24
Change in physical activity energy expenditure score as measured by Recent Physical Activity Questionnaire (Metabolic Equivalent of Task hours/day) | Change from Baseline to Week 12 and to Week 24
Change in Gut microbiota composition as measured by fecal microbial alpha-diversity, beta diversity and taxa abundances using metagenomic approach | Change from Baseline to Week 24
Change in Gut microbiota function as measured by fecal microbial pathways abundances using metagenomic approach | Change from Baseline to Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No